CLINICAL TRIAL: NCT01828164
Title: The Effect of Ultrasound on Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SmileSonica Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-0018-0031-0041; 197850 (Other: Health Canada)
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Malocclusion
Keywords: Orthodontics; Braces; Tooth
MeSH Terms: conditions — Malocclusion | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): 20 minutes per day of ultrasound treatment on the active side of the device. The device consists of a mouth guard type device with transducers embedded in the mouth guard. In the split mouth design, the treatment arm consist of the side of the mouth with the transducers activated.
  Interventions: Device: Ultrasound
- Control Arm (Sham Comparator): The transducers are not activated on the control side of the device.The subjects wear the device for 20 minutes per day for the duration of the study. The device consists of a mouth guard type device with transducers embedded in the mouth guard. In the split mouth design, the control arm consist of the side of the mouth with the transducers deactivated.
  Interventions: Device: Sham comparator

INTERVENTIONS:
Device: Ultrasound — The Aevo System™ is an ultrasound emitting dental device.
  Other Names: Aevo System.
  Arms: Treatment Arm
Device: Sham comparator — Ultrasound not activated in the comparator side of the device.20 minutes per day of ultrasound treatment on the active side of the device. The device consists of a mouth guard type device with transducers embedded in the mouth guard. In the split mouth design, the treatment arm consist of the side of the mouth with the transducers activated while the comparator arm has the transducers deactivated.
  Arms: Control Arm

SUMMARY:
To study whether or not the Aevo System™ medical device enhances the rate of tooth movement in human subjects who use orthodontic braces.

DETAILED DESCRIPTION:
The study will involve comparing the effects of tooth movement with and without ultrasound treatment in a split mouth design. Treatment will consist of using the Aevo System™ device for one 20 minute period per day for the duration of the trial (up to 24 weeks). Tooth position measurements will be taken from eligible patients prior to commencing usage of the study device. Follow-up visits will be scheduled for intra-oral clinical measurements and to take full-arch impressions. The Aevo System™ consists of an ultrasound emitting mouthpiece which is wire connected to an external handheld device. The mouthpiece is placed over the teeth and over the braces every day for 20 minutes in order to deliver the therapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will qualify for entry into the study:

1. Scheduled to receive orthodontic treatment or in early stage of orthodontic treatment
2. Minimum of 3 mm of extraction space (on both sides of a dental arch) to be closed either by distal movement of all 6 anterior teeth from canine to canine or by distal movement of the canines.
3. Available for follow-up visits.
4. Willing and able to sign written informed consent.
5. Healthy.
6. Has permanent dentition and between the ages of 12 and 40.
7. Good oral hygiene and compliance

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Any compromised medical or dental condition that prevents the subject from participating in the trial or using the medical device.
2. Any implanted assistive devices.
3. Currently involved in any other study.
4. Lives significantly outside the clinical trial site.
5. Use of bisphosphonates.
6. Pregnant females .

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek El-Bialy, PhD, FRCD(C), Principal Investigator — University of Alberta, Department of Dentistry; Kevin L Knowlton, DDS, Principal Investigator — Faculty of Dentistry, University of Toronto; Bryan D Tompson, DDS, FRCD(C), Principal Investigator — Faculty of Dentistry, University of Toronto; Terry Carlyle, DDS, MS, Principal Investigator — Strathcona Orthodontics, Edmonton; William Wiltshire, BChD, ChD, Principal Investigator — Faculty of Dentistry, University of Manitoba; Tim Dumore, DMD, BS, MS, Principal Investigator — Dr. Dumore and Team Orthodontics, Winnipeg
Locations (5):
- Canada (5):
  - Site 3: Strathcona Orthodontics Clinic, Edmonton, Alberta
  - Site 1: University of Alberta, Facilty of Dentistry, Edmonton, Alberta
  - Site 4: Faculty of Dentistry, University of Manitoba, Winnipeg, Manitoba
  - Site 5: Dr. Dumore and Team Orthodontics, Winnipeg, Manitoba
  - Site 2: Faculty of Dentistry, University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 subjects did not meet inclusion criteria after enrollment. For this reason, 60 subjects were enrolled but only 49 entered the participant flow.
Groups:
- All Study Participants: As per split mouth design, one side of the mouth received treatment while the other side of the mouth served as the control. In this design, each subject was both treated and served as control.
Period: Overall Study
Arm/Group | All Study Participants
Started | 49 (11 out of 60 subjects did not meet inclusion criteria after enrollment.)
Completed | 32
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.4 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13
Region of Enrollment [Number; unit: participants]
  Canada | 49

OUTCOME MEASURES:

1. Primary Outcome: Rate of Tooth Movement
Description: The weekly rate of tooth movement (mm/week) as compared between the treated side and the control side.
Time Frame: 24 weeks or until the extraction space was closed (whichever came first)
Population: As per approved protocol, only subjects who completed the study with device usage compliance of 67% or higher and with functional devices were evaluated.
Measure: Mean (Standard Deviation); unit: mm/week
Groups:
- Treatment Arm: The side of the mouth that received treatment. As per split mouth design, one side received treatment while the other side served as the control. In this design, each subject was both treated and served as control.
- Control Arm: The side of the mouth that was the control. As per split mouth design, one side received treatment while the other side served as the control. In this design, each subject was both treated and served as control.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 17 | 17
mm/week | 0.266 (0.0927) | 0.232 (0.0855)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Superiority or Other; p = 0.0164, t-test, 1 sided; Percent Change = 29.0 — Percent change in tooth movement rate on the treatment side as compared to the control side

2. Secondary Outcome: Rate of Root Resorption
Description: The weekly rate of tooth root resorption (mm/week) as compared between the treated side and the control side.
Time Frame: 24 weeks or until the extraction space was closed (whichever came first)
Population: Subjects who completed the study with device usage compliance of 67% or higher and with functional devices were evaluated. Only subjects with CBCT images were used.
Measure: Mean (Standard Deviation); unit: mm/week
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 13 | 13
mm/week | 0.0092 (0.0226) | 0.0241 (0.0223)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Superiority or Other; p = 0.0423, t-test, 1 sided; Percent change = 220.8 — Percent change in root resorption rate on the control side as compared to the treatment side

3. Secondary Outcome: Discomfort
Description: Average measured level of subject discomfort or pain. The Participant Pain Reporting Scale is used to assess the amount of pain on a 10 point scale. On the 10 point scale, 1 represents the least amount of pain and 10 represents the most amount of pain.
Time Frame: 24 weeks or until the extraction space was closed (whichever came first)
Population: Subjects who completed the study with device usage compliance of 67% or higher.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment Arm: The side of the mouth that received treatment. As per split mouth design, one side of the mouth received treatment while the other side of the mouth served as the control. In this design, each subject was both treated and served as control.
- Control Arm: The side of the mouth that was the control. As per split mouth design, one side of the mouth received treatment while the other side of the mouth served as the control. In this design, each subject was both treated and served as control.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 24 | 24
units on a scale | 1.990 (2.030) | 2.000 (1.713)
Statistical Analysis 1: Comparison: Treatment Arm vs Control Arm; Test type: Non-Inferiority — 1 point on the 10-point pain scale was used as the non-inferiority margin; p < 0.001, Bootstrapped mean difference; This test bootstrapped the mean difference (Treatment Arm - Control Arm) less 1, the non-inferiority margin, 1000 times

ADVERSE EVENTS:
Time Frame: The duration of the study, up to 24 weeks.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less